CLINICAL TRIAL: NCT02921945
Title: A Multi-center, Phase III, Non-controlled, Open-label Trial to Evaluate the Safety and Efficacy of SCT800 for On-demand Treatment in Previously Treated Patients With Hemophilia A
Brief Title: Efficacy and Safety Study of SCT800 for On-demand Treatment With in Patients With Hemophilia A
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT800HA3
Record Dates: First submitted 2016-09-28; First posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCT800 (Experimental)
  Interventions: Biological: SCT800

INTERVENTIONS:
Biological: SCT800 — recombinant human coagulation factor VIII

SUMMARY:
In this trial safety and efficacy of SCT800 (B-domain deleted recombinant factor VIII) is being evaluated in 50 subjects, 12 to 65 years of age, with moderate to severe Hemophilia A. These subjects will receive open label treatment with SCT800 for approximately 6 months for on-demand treatment.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 65 years old;
* The activity of the coagulation factor VIII (FVIII:C) ≤5%, and was previously treated with FVIII concentrate(s) for a minimum of 50 exposure days (EDs) prior to study entry
* Bleeding state need to be treated with FVIII;
* Negative assays for FVIII inhibitors (<0.6 BU/mL);
* The platelet count is normal；
* Normal prothrombin time or INR ≤1.5；
* Given informed consent

Exclusion Criteria:

* Hypersensitivity to recombinant coagulation factor VIII concentrate or any of the excipients ;allergic to heterologous proteins (e.g. murine, bovine or hamster origin);
* Family history or history of FVIII inhibitors (≥0.6 Bethesda Units [BU] mL-1);
* Received an infusion of any FVIII for on-demand therapy or prophylaxis within 4 days prior to study entry (including rFVIII, plasma-derived factor VIII [pdFVIII], cryoprecipitate and whole blood);
* Significant hepatic or renal impairment (ALT and AST ≥2×ULN; BUN and Cr≥2×ULN);
* HIV seropositive;
* Abnormal hemostasis from causes other than hemophilia A；
* Patients with severe heart disease, including myocardial infarction, heart failure (III or higher level);
* Patients who received any anticoagulant or antiplatelet therapy within one week (including NSAIDs) or need to receive an anticoagulant or antiplatelet therapy during the period of clinical trials;
* Alcoholism, drug abuse, mental disorders and mental retardation;
* Elective surgery planned during the process of study;
* Patients who previously participated in the other clinical trials prior to study entry;
* The patient or parent/legal guardian is unable or unwilling to sign an informed consent form or to comply with the requirements of clinical protocol;
* Other conditions confirmed by the researchers, resulting in that patients are unable to benefit from clinical observation;

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Incremental Recovery (K-value) | 1hour after the end of the infusion
  One-stage aPTT Assay

SECONDARY OUTCOMES:
Haemostatic effect of SCT800 evaluated according to a predefined four grade scale: excellent, good, moderate, or no response | Up to 6 months
The incidence rate of FVIII inhibitors (≥0.6 BU) | Up to 6 months
The number of infusions of SCT800 required per bleeding episode | Up to 6 months
Actual consumption of SCT800 (IU/Kg/bleed) | Up to 6 months
AEs related to SCT800 during the clinical study | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xielan Zhao, PhD, Principal Investigator — Xiangya Hospital of Centre-South University, Changsha, China
Locations (1):
- Xiangya Hospital of Centre-South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No